CLINICAL TRIAL: NCT01194492
Title: Albumin Kinetics in Generalized Inflammation - an Exploratory Study on Patients Before and After Major Abdominal Surgery
Brief Title: Albumin Kinetics in Generalized Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ake Norberg, MD PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-018529-21
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Major Abdominal Surgery
Keywords: plasma albumin; inflammatory reaction; systemic inflammatory response syndrome
MeSH Terms: conditions — Inflammation; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Albumin kinetics (Other)
  Interventions: Radiation: Albumin transcapillary escape rate (125I-albumin)

INTERVENTIONS:
Radiation: Albumin transcapillary escape rate (125I-albumin) — Repeated measure by injection of 0.1 megabecquerel and 0.3 megabecquerel of 125-iodine labeled albumin before surgery and 2 days after surgery, respectively.
  Other Names: SERALB-125

SUMMARY:
The purpose of this study is to determine whether the kinetics of endogenous albumin is altered by the generalized inflammation caused by major abdominal surgery.

DETAILED DESCRIPTION:
Albumin infusions have been used for expansion of the plasma volume for more than 60 years, not only in the operating room, but also in trauma and sepsis. However, there is an ongoing debate whether albumin is good or bad for the patient compared to other intravenous fluids, in different situations. Our research program aims at exploring this issue, starting by describing how the body handles the endogenous albumin in connection with severe inflammation. The final goal is to improve fluid treatment for these patients.

Plasma albumin is often decreased in inflammation. However, the underlying mechanisms are not well described. Two aspects of albumin kinetics will be covered in this study by measurements immediately before and two days after major abdominal surgery, that will serve as a model for generalized inflammation. Albumin fractional synthesis rate will be determined by the incorporation of deuterium labelled phenylalanine into plasma albumin. Albumin distribution will be measured as transcapillary escape rate of radioiodinated albumin. By assessment of P-albumin and plasma volume it will be possible to calculate albumin absolute rate of synthesis and albumin absolute flux from the central compartment, respectively.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patients planned for major abdominal surgery, pancreatic
* age ≥ 40 years

Exclusion Criteria:

* pregnant or lactating patients
* planned peri-operative infusions of albumin or plasma
* S-creatinine > 110 mmol/L
* allergy against iodine
* other conditions preventing the subject from participating in the study, as judged by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in albumin transcapillary escape rate | 2 days
  Transcapillary escape rate is measured as the rate of decrease of 125I-albumin in plasma over 90 min. The assessment is performed twice, immediately before surgery and in the second post-operative day, respectively.
Change from baseline in albumin synthesis rate | 2 days

SECONDARY OUTCOMES:
Changes from baseline in markers of inflammation (heart rate, respiratory rate, body temperature, Blood leukocyte count, and P-CRP) | 2 days
  The markers of inflammation is measured twice in each patient, immediately before and two days after surgery, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Sigridur Kalman, MD, Ass Prof, Study Chair — Karolinska Institutet, Institution of Clinical Science Intervention and Technology, Dept of Anesthesiology
Locations (1):
- Karolinska University Hosptial, Huddinge, Stockholm, Sweden

REFERENCES:
- [Result] Norberg A, Rooyackers O, Segersvard R, Wernerman J. Albumin Kinetics in Patients Undergoing Major Abdominal Surgery. PLoS One. 2015 Aug 27;10(8):e0136371. doi: 10.1371/journal.pone.0136371. eCollection 2015. PMID 26313170